CLINICAL TRIAL: NCT03094598
Title: The INFO-I Trial: A Randomised Trial Assessing the Impact of Written Information on Outpatients' Knowledge About and Attitude Toward Randomised Clinical Trials
Brief Title: Outpatients' Knowledge About and Attitude Toward Randomised Clinical Trials
Acronym: INFO-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Collaborators: The Info Trial Group (Other); Charlotte Behnke (Unknown); Pia Caspersen (Unknown); Dorte Fischer (Unknown); Rolf I. Hansen (Unknown); Karin Jensen (Unknown); Birthe Klarskov (Unknown); Lars K. Møller (Unknown); Kirsten Obel (Unknown); Sten N. Rasmussen (Unknown); Pia Munkholm (Unknown); Ju-ri Rumessen (Unknown); Stig Sonne-Holm (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Protokol: 1996-10-31/KK.df; 1996-DP-18-RKF-3-INFO-I (Other: CTU)
Record Dates: First submitted 2016-08-25; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Ambulatory Patients in the Dep. of Medical Gastroenterology; Ambulatory Patients in the Dep. of Gynecology; Ambulatory Patients in the Dep. of Orthopedic Surgery; Ambulatory Patients in the Dep. of Urology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): No intervention
- Leaflet (Experimental): The leaflet is based on information and journalism theories, paying attention primarily to reader appeal and readability.
  Interventions: Other: Leaflet
- Brochure (Experimental): The brochure is based on practical communication experience, focusing primarily on logical composition and presentation of condensed information.
  Interventions: Other: Brochure
- Booklet (Experimental): The booklet is also based on practical communication experience, but give more elaborate explanations.
  Interventions: Other: Booklet

INTERVENTIONS:
Other: Leaflet — The length is 1.5 A4 pages, Flesch's Reading Ease Score (RES) is 57 (fairly difficult, comparable to a quality magazine), and Human Interest Score (HIS) is 37 (interesting, comparable to a digest magazine).
  Arms: Leaflet
Other: Brochure — The length is 2.5 A4 pages, RES is 43 (difficult, comparable to an academic magazine), and HIS is 25 (interesting, comparable to a digest magazine).
  Arms: Brochure
Other: Booklet — The length is 12 A4 pages, RES is 11 (very difficult, comparable to a scientific magazine), and HIS is 22 (mildly interesting, comparable to a trade magazine).
  Arms: Booklet

SUMMARY:
The purpose of this study is to investigate the knowledge about randomised clinical trials and the attitude towards clinical research among Danish outpatients. The INFO Trial was designed as a randomised, parallel group, observer-blinded trial comparing three types of written information (a leaflet, a brochure, and a booklet) to each other and to a no intervention group.

DETAILED DESCRIPTION:
To improve the patient education process in clinical research, three information materials describing general aspects of design and conduct of randomised clinical trials were developed. The materials varied in length, reading ability level, and reader appeal. Their influence on knowledge about and attitude toward randomised clinical trials was assessed in a randomised, parallel group, evaluator-blinded trial among 415 outpatients recruited from four departments at a university hospital in Copenhagen. The patients were randomised to the following groups: control (no intervention), leaflet, brochure, or booklet in a 1:1:1:1 ratio. Knowledge (KN) was assessed by a 17-item multiple-choice questionnaire and attitude (AT) was assessed by a 32-item Likert questionnaire at entry and 2 weeks after the intervention. The interventions and the questionnaires were pilot tested and power calculations were performed.

Assessment of scales for knowledge and attitudes was performed using Rasch analysis and Cronbach 's alpha. Associations between demographic variables, knowledge score and attitude score were examined using analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* Ability to read and understand Danish and written informed consent.

Exclusion Criteria:

* Patients under 18 years of age and patients enrolled in another clinical trial on the same day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 1996-10; Primary Completion 1996-12 (Actual); Study Completion 1996-12 (Actual)

PRIMARY OUTCOMES:
Knowledge (KN) scores | 2 weeks
  Change in knowledge (KN) scores scores between entry and follow-up.

SECONDARY OUTCOMES:
Attitude (AT) (total) scores | 2 weeks
  Change in attitude (AT) (total) scores between entry and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Krogsgaard, MD, Principal Investigator — Copenhagen Trial Unit - Centre for Intervention Research, Denmark
Locations (2):
- Denmark (2):
  - Copenhagen Trial Unit, Centre for clinical intervention research, Copenhagen
  - Hvidovre University Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No
No plan for data sharing

REFERENCES:
- [Result] Kruse AY, Kjaergard LL, Krogsgaard K, Gluud C, Mortensen EL, Gottschau A, Bjerg AM. A randomized trial assessing the impact of written information on outpatients' knowledge about and attitude toward randomized clinical trials. The INFO trial group. Control Clin Trials. 2000 Jun;21(3):223-40. doi: 10.1016/s0197-2456(00)00048-9. PMID 10822120
- [Result] Kjaergaard LL, Kruse AY, Krogsgaard K, Gluud CN, Mortensen EL, Gottschau A, Bjerg AM. Outpatients' knowledge about and attitude towards clinical research and randomized clinical trials. The INFO Trial Group. Dan Med Bull. 1998 Sep;45(4):439-43. PMID 9777295